CLINICAL TRIAL: NCT06278883
Title: Deploying a Genomic-medicine Risk Assessment Model for Diverse Primary Care Populations and Settings
Brief Title: Genomic Medicine Risk Assessment Care for Everyone - Implementation Phase
Acronym: GRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00115007; R01HG011794 (NIH)
Record Dates: First submitted 2024-01-31; First posted 2024-02-26 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Diseases; Cancer; Liver Diseases; Hyperthermia
Keywords: implementation science; risk assessment; genetics; cascade screening; family history; hereditary conditions; genetic testing; genetic counselling
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Liver Diseases; Hyperthermia

STUDY DESIGN:
Intervention Model Description: Everyone who consents is enrolled in the risk assessment pipeline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Risk assessment pipeline
  Interventions: Behavioral: Disease Risk Assessment

INTERVENTIONS:
Behavioral: Disease Risk Assessment — Undergo personal and family history-based risk assessment and make recommendations for managing risk.

SUMMARY:
The "Genomic medicine Risk Assessment Care for Everyone" (GRACE)" intervention project will develop a scalable end-to-end solution for risk assessment and management that meets the needs of those populations living in low resource settings. The long-term goal is to increase access to and uptake of risk-informed evidence-based guidelines that will improve population health through better patient outcomes, higher quality of life, and decreased costs. The three primary aims are:

Aim 1: Develop a scalable implementation framework that guides each unique clinical setting, including low resource settings, in deploying GRACE effectively for the needs of their patients and providers.

Aim 2: Facilitate the potential for genomic medicine to promote population health by broadening access to and uptake of genomic risk assessment by the general population through a pragmatic implementation-effectiveness trial of GRACE.

Aim 3: Reduce health disparities related to genomic medicine by allowing individual adaption of GRACE to suit their level of resources, education, and access within a pragmatic implementation-effectiveness trial.

Three sets of participants will be engaged: patients (n=750), providers (n=25), and family members of "probands" (i.e., patients that have a genetic change that increases risk, n~500).

Patient participants will be asked to complete a baseline survey, enter their family health history information into MeTree (a family health history web-based platform) and complete a survey about their experience using the platform. Subsequent study procedures will depend on: 1) the results of their MeTree risk evaluation, 2) their acceptance/declination of genetic testing (for those categorized as needing testing by MeTree), and 3) the results of the test (for those accepting testing).

Provider participants will be providers who are the primary care physicians treating one or more patients enrolled in the patient participant group. Providers will be notified on a patient by patient basis once the patient participant under their care has complete the risk assessment process and the risk report is available from MeTree. At study completion, provider participants will be asked to complete a survey about their demographics, practice, and experiences with the study.

Blood relatives of the probands who are identified by the proband as open to engaging with the study will be contacted and offered genetic counseling and genetic testing.

DETAILED DESCRIPTION:
The "Genomic medicine Risk Assessment Care for Everyone" (GRACE)" project will define, deploy and evaluate a new care delivery model. Specifically, the GRACE project will develop a scalable end-to-end solution for risk assessment and management that meets the needs of those populations living in low resource settings. The long-term goal is to increase access to and uptake of risk-informed evidence-based guidelines that will improve population health through better patient outcomes, higher quality of life, and decreased costs. The central hypothesis is that combining a Family Health History (FHH) -driven risk assessment tool (in this case MeTree), family engagement, and a genetic testing delivery system, will create a solution that engages and increases the proportion of diverse patients who are identified as at increased risk, who undergo testing, and, when appropriate, who initiate cascade genetic testing among relatives. The three primary aims are:

Aim 1: Develop a scalable implementation framework that guides each unique clinical setting, including low resource settings, in deploying GRACE effectively for the needs of their patients and providers.

Aim 2: Facilitate the potential for genomic medicine to promote population health by broadening access to and uptake of genomic risk assessment by the general population through a pragmatic implementation-effectiveness trial of GRACE.

Aim 3: Reduce health disparities related to genomic medicine by allowing individual adaption of GRACE to suit their level of resources, education, and access within a pragmatic implementation-effectiveness trial.

This trial is a cluster step wedge design, meaning that while the trial will ultimately be implemented in five family medicine clinics at the University of Florida Health System, it will be implemented in only one clinic at a time.

Briefly, when one clinic has completed enrollment of the target number of patients (n=150) and providers (n=3-5), then the investigators will advance to enrolling patients and providers in the next clinic. That is, the investigators will not wait until blood relatives of the probands are recruited before moving to the next clinic. Finally, in the spirit of implementation science, the investigators will evaluate the lessons learned, barriers and facilitators from each clinic and use this knowledge so that the next clinic will benefit from the experiences of the previous ones.

Three sets of participants will be engaged: patients (n=750), providers (n=25), and family members of "probands" (i.e., patients that have a genetic change that increases risk, n~500).

Patient participants will be asked to complete a baseline survey, enter their family health history information into MeTree (a family health history web-based platform) and complete a survey about their experience using the platform. Once data entry in MeTree is complete, all participants will be able to view and download a personalized patient report within the platform outlining their familial and genetic/hereditary risk status that includes medical conditions according to current evidence-based guidelines. The report will indicate whether the participant has a) population-level risk (also referred to as not at high risk) suggesting nothing different needs to be done with their preventive care, b) familial risk (suggesting a change in care, but no need for genetic testing), or c) hereditary risk (suggesting a need for genetic testing and that they might also meet criteria for changes in preventive care).

Subsequent study procedures will depend on: 1) the results of their MeTree risk evaluation, 2) their acceptance/declination of genetic testing (for those categorized as needing testing by MeTree), and 3) the results of the test (for those accepting testing). Based on these three factors, patients will fall into one of five groups (see below).

GROUP 1: Not at High Risk, No Testing Recommended (n~400).

GROUP 2: Familial Risk, Genetic Testing not recommended, clinical care recommended (n~100).

GROUP 3: Genetic Risk, Testing Recommended, Testing Declined, (n~60)

GROUP 4: Genetic Risk, Testing Recommended, Testing Accepted, Negative Test Result (n~140)

GROUP 5: Genetic Risk, Testing Recommended, Testing Accepted, Positive Test Result (n~50)

Participants in Groups 1 and 2 will be asked to complete a survey to assess their reflections on their risk assessments. After completing this survey, they will have completed all study activities.

Study procedures for participants in Groups 3-5 (those identified as having a hereditary risk) will be determined by the number of diseases they are at risk for according the MeTree risk assessment.

* Patient participants identified to be at genetic risk of multiple diseases under study (i.e. certain cancers and/or cardiovascular and/or liver diseases) will be contacted a genetic counselor who will provide clinical pre-test genetic counseling, which is part of normal clinical care for genetic counseling. The genetic counselor will offer these patient participants genetic testing, which they can decline. Of note, their acceptance/declination and the results of the test (for those who accept testing) will determine if they are in Group 3, 4 or 5).
* Patient participants identified to be at genetic risk for a single disease under study (i.e. certain cancer, cardiovascular, or liver diseases) will be provided with access a virtual Genetic Information Assistant (GIA) chatbot that is specific to their risk category. They will also be invited to view a short video describing the purpose of the chatbot. Once in the chatbot, participants will be offered genetic counseling through GIA or the option to obtain clinical genetic counseling through a study genetic counselor. If the participant does not access the GIA chatbot within 2 weeks after having access, a team member will contact the participant to offer support for GIA or genetic counseling with a study genetic counselor.
* Patient participants who decline to undergo genetic counseling or testing (Group 3) will be asked why they elected not to receive genetic counseling or genetic testing. They will also be asked to complete a survey about their experience with the study. After completing this survey, participants in Group 3 will have completed the study.
* Patient participants who agree to undergo genetic counseling and genetic testing will receive a saliva collection test kit for genetic testing to mail to Invitae, the company that will assist with genetic testing. A mobile phlebotomy unit will also be available and can be deployed to collect blood for genetic testing, if preferred/needed.

  * For patient participants whose genetic test result is negative (Group 4), suggesting no evidence of a genetic change that increases risk of diseases under study, results will be returned by GIA if they had pre-test counseling by GIA or by a study genetic counselor if they had pre-test counseling by a study genetic counselor. After the genetic test results are returned, participants in this group will be asked to complete a survey about their experience with genetic counseling. After completing this survey, participants in Group 4 will have completed the study.
  * For patient participants whose genetic test result is positive (Group 5), suggesting evidence of a genetic change that increases risk of one or more of the diseases under study, a study genetic counselor will return their results and encourage them to share their results with blood-related family members, as is standard practice during routine return of result counseling for those with a positive finding. The study genetic counselor will give the patient participant a standard family member letter to help facilitate sharing of information and cascade screening. Participants will be asked to complete a post genetic counseling/genetic testing survey, which includes questions regarding whether they shared information with blood-related family members, with whom, and contact information for adult blood-related family members who have indicated they are receptive to direct contact by the study team about cascade screening. After completing this survey, these participants will have completed the study.

Blood relatives of the probands who are identified by the proband as open to engaging with the study will be contacted. If they are a resident in North Carolina, Florida, South Carolina, West Virginia, New York, Maine, Texas, Mississippi, Missouri, Kansas, Colorado, Arizona, or Alaska, they will be offered genetic counseling with study genetic counselor. GRACE study genetic counselors are licensed in both Florida and North Carolina. The other states listed do not require in-state licensure for genetic counseling. If the blood relative is not a resident in one of these states, a study team member will provide recommendations for genetic counseling and testing, including through a) University of Pennsylvania's eREACH 2.0 study where participants can receive free genetic counseling and family variant testing regardless of state of residence, b) Genome Medical (a company associated with Invitae who will do the proband's genetic testing), who offers pre- and post-test genetic counseling sessions for $199. The family variant testing itself is free through Invitae, and c) the National Society of Genetic Counselors "Find a Genetic Counselor" resource. Approximately 3 months after consenting to participate in the study, blood relatives will receive a survey about their perceptions and experience with the direct contact process, what the patient participant shared with them prior to contact by the study team member, if they have been given the family member letter, what information they found helpful, if they had any concerns about the process, what information helped them decide whether to get counseling, what their decision was, what information was helpful in making this decision, and what factors informed their decision to get testing or not. After completing the survey, blood relatives will have completed the study.

Provider participants will be providers who are the primary care physicians treating one or more patients enrolled in the patient participant group. Providers will be notified on a patient by patient basis once the patient participant under their care has complete the risk assessment process and the risk report is available from MeTree. Providers will be notified via EPIC messaging or an alert that their patient has a MeTree clinical decision support report available in the patient's electronic medical record. Whether the provider reviews the risk assessment or changes patient care based on risk assessment recommendations is part of standard clinical care and will be evaluated as a study outcome. Notification will also occur when a patient declines genetic counseling, declines genetic testing, or has completed genetic testing return of results. Eligibility for genetic counseling will be noted in the medical record if a patient declines. If the patient undergoes genetic counseling, as is standard of care, genetic counseling recommendations for testing, and testing outcomes will also be documented in the medical record. When all patient participants in a clinic have completed all study procedures, provider participants will be asked to complete a survey, which will include questions about their demographics, practice, and experiences with the study. After completing the survey, provider participants will have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Receiving primary medical care in one of the 5 participating clinics
* Age 18 years or older
* Able to read and communicate in English
* Able to provide written and verbal informed consent
* Willing to use the Internet

Exclusion Criteria:

* Anyone not meeting inclusion criteria
* Previous genetic counseling and/or previous hereditary panel testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Reach of genomic risk assessment | at study completion, expected 1 year from study start
  The number of participants completing MeTree relative to the number of participants who consented to the study.
Utility of genomic risk assessment | at study completion, expected 1 year from study start
  The number of participants newly identified as at increased risk for familial and/or heritable conditions warranting genetic counseling and/or genetic testing.
Uptake of genetic counseling risk recommendations by the participant | at study completion, expected 1 year from study start
  The number of participants who complete genetic counseling/the number of participants who are recommended for genetic counseling.
Uptake of genetic testing recommendations by the provider | at study completion, expected 1 year from study start
  The number of participants who undergo genetic testing/the number of participants recommended for genetic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Orlando, MD, Principal Investigator — Duke University; Alexander S Parker, PhD, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - UF Health Family Medicine - Lem Turner, Jacksonville, Florida
  - UF Health Family Medicine - Commonwealth, Jacksonville, Florida
  - UF Health Augustine Oaks, Jacksonville, Florida
  - UF Health Oakleaf, Orange Park, Florida

IPD SHARING:
Plan to Share IPD: Yes
Diagnostic genomic testing data will be deposited in an appropriate NIH data repository once the study team makes a final determination (e.g., dbGaP). Additional data documentation and de-identified data will be deposited along with phenotypic data, which includes demographics, family history of diseases collected through the MeTree program, and diagnosis, consistent with applicable laws and regulations. The study investigators will comply with the NIH genome-wide association studies (GWAS) Policy and the funding IC's existing policies on sharing data on specified disease genetics to include secondary analysis of data resulting from a genome wide association study through the repository. Meta-analysis data and associated phenotypic data, along with data content, format, and organization, will be available. Submitted data will conform to relevant data and terminology standards.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available 6 months after publication and be available indefinitely.
Access Criteria: The data will be deposited in an NIH data repository (e.g., dbGaP) for access by others that conforms to the following criteria: 1) used solely for research purposes, 2) properly acknowledged in resulting publications, 3) kept confidential and inaccessible to third parties, and 4) destroyed or returned after analyses are completed. Additionally, users must agree not to use data to identify individual participants.

DOCUMENTS (1):
  • Informed Consent Form (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT06278883/ICF_000.pdf